CLINICAL TRIAL: NCT06875271
Title: Inclinometer Assessment of Seated Shoulder Position Sense: Intra- and Inter-Rater Reliability and Validity
Brief Title: Inclinometer Reliability in Seated Shoulder Position Sense Assessment
Status: Active, not recruiting | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FSM PRH schoulder
Record Dates: First submitted 2025-02-24; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Position Sense

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Inclinometer Assessment of Seated Shoulder Position Sense: Intra- and Inter-Rater Reliability and Validity

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants aged 18-60 with no current or past shoulder injury, trauma, or pain.

Exclusion Criteria:

* Pain in the upper extremity or neck
* Limited range of motion in the upper extremity joints
* Any history of upper extremity, cervical, or cranial injury
* Regular involvement in a sport or occupation that requires frequent overhead shoulder movements
* Performing strenuous exercise within 24 hours prior to the assessment
* Consumption of alcohol and/or illicit substances within 24 hours prior to the assessment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy participants aged 18-60 with no current or past shoulder injury, trauma, or pain.
Sampling Method: Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Position Sense | 1 day
  This study is an observational, cross-sectional investigation conducted to evaluate shoulder joint position sense (JPS) in healthy volunteers. It aims to assess the reliability of JPS measurements performed in a seated position using a digital inclinometer.
  Experimental Procedure:
  In this study, shoulder joint position sense (JPS) measurements will be conducted in a seated position using a digital inclinometer.
  Test Protocol:
  Participants will be asked to reproduce three different shoulder flexion and abduction angles:
  Low range: 55° ± 5° Middle range: 90° ± 5° High range: 125° ± 5° Participants will also be asked to reproduce a 20° ± 5° shoulder internal rotation (IR) and external rotation (ER) angle in the horizontal plane.
  After raising their arm to a randomly determined angle and holding it for a few seconds, they will be instructed to return to the starting position.
  They will then be asked to reproduce the angle they remember.

CONTACTS AND LOCATIONS:
Overall Officials: pmr specialist, Principal Investigator — Liv hospital vadistanbul
Locations (1):
- Liv hospital Vadistanbul, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP